CLINICAL TRIAL: NCT05144269
Title: Investigation of the Effects of Multimodal Exercise-Based Telerehabilitation on Psychosocial Factors in Postpartum Women
Brief Title: Telerehabilitation in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Yaprak Cetin, PT, Asst, Prof, PhD, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-400
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Postpartum Women; Telerehabilitation
Keywords: Postpartum; Depression; Physical activity; Pilates; Telerehabilitasyon
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal exercises group (Experimental): Multimodal exercise-based telerehabilitation will be implemented with video conference method. For telerehabilitation, a program including pilates, breathing, progressive relaxation training, posture and pelvic floor strengthening exercises was created. Sessions consist of 45 minutes. Telerehabilitation will take place 2 days a week for 8 weeks.
  Interventions: Other: Multimodal exercises
- Education group (No Intervention): 30 minutes of training will be given about postpartum and exercises. As exercise, only aerobic walking exercise, which can be started for 15 minutes a day and 3 days a week according to the guide, gradually increasing, up to 30 minutes and up to 4 days a week will be applied. There will also be a warm-up and a cool-down period before the walking exercise. *Exercise intensity is determined in the 12-14 score range according to the Borg Scale, and how to apply it will be explained.

INTERVENTIONS:
Other: Multimodal exercises — Telehabilitation including pilates, breathing, progressive relaxation training, posture and pelvic floor strengthening exercises
  Arms: Multimodal exercises group

SUMMARY:
Postpartum is a transitional period in which physical, social and emotional changes take place in the women. Especially the difficulty of psychological and physiological changes can be associated with deterioration in the women's health. Exercise support programs given to postpartum women have been shown to contribute to physical, mental and social well-being. Statistically significant improvements were found in depression and anxiety symptoms, energy and fatigue parameters, and general health regarding the effects of exercise on mental health in pregnant and postpartum women. The recommendation of the American Association of Obstetricians and Gynecologists (ACOG) is that women start physical activity as soon as they are medically or obstetrically safe. It is stated that they can be included in the exercise programs as soon as possible if it is a normal delivery, and after the 6th week, except for certain exercises if it is a cesarean section. Literature mentioned that exercise studies with postpartum women are insufficient. These mostly focused on the postpartum period and women who had a cesarean section were excluded. In their studies comparing the clinical and virtual environment; Although there is no statistical difference, there are studies showing that it is superior. To the best knowledge, there were no studies on postpartum telerehabilitation. Literature with a multidimensional approach in line with the recommendations of the guidelines were also limited.

DETAILED DESCRIPTION:
This study is a randomized controlled trial aiming to examine the improvement in psychosocial status and physical activity in postpartum women after 8 weeks of multimodal exercise-based telerehabilitation. Two groups will be formed, namely the intervention group and the training group.

Multimodal exercise-based telerehabilitation will be applied to the intervention group by an experienced physiotherapist in 45-minute sessions, 2 days a week, for 8 weeks; Postpartum and exercise related training will be given and they will be asked to walk gradually increasing aerobic exercises. All interventions are common except for the control group telerehabilitation. Women will be evaluated before and after the study. 'Edinburgh Postpartum Depression Scale (EPDS)', 'Fatigue Severity Scale (FSS)', 'Pittsburgh Sleep Quality Index (PUKI), 'World Health Organization Lifestyle' for depression, fatigue, sleep, quality of life, physical activity and mental health in evaluations. World Health Organization Quality of Life Scale (WHOQOL-BREF)', 'Kaiser Physical Activity Questionnaire (KFAA)', 'Short Symptom Inventory' will be used.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum between 6-12 weeks
* giving birth to a healthy baby
* Having technological devices that can be connected online via video conferencing,
* women who can use technological devices to connect

Exclusion Criteria:

* Multiple pregnancy,
* Having other diseases that will affect their functions,
* Having a problem related to the musculoskeletal system (such as abdominal hernia) that will prevent exercise,
* having neurological, rheumatic disease
* having chronic pain
* Diastasis recti distance greater than 2 cm,
* Women whose babies were hospitalized during the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in the postpartum period who have just given birth
Enrollment: 58 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postpartum Depression Scale | 2 months
  The Edinburgh Postpartum Depression Scale, developed by Cox and Holden, is used to determine the risk of depression in the postpartum period and to measure the change in level and severity. The scale is a self-assessment scale consisting of 10 questions in 4-point Likert type. The scores obtained from the scale vary between 0-30. The cut-off point is 13 and those who score 13 and above are considered to have depression risk/suspicion.
Kaiser Physical Activity Questionnaire | 2 months
  It was adapted from the Baecke Physical Activity Questionnaire to measure physical activity in women. In the scale, both how often the activities are done and how much time is spent on that activity are questioned. The survey consists of 38 questions in total. The questions in the survey are grouped under four main headings: "housework/care", "occupational", "active life", "sports and exercise". There are 11, 8, 4 and 15 questions in these categories, respectively. The questions are scored from 1 to 5. The scores of each category are averaged. It is then multiplied by the frequency, duration and MET value and summed up on all activities. The MET values of 3.5, 5 and 7, respectively, were used to represent the average MET values of activity in each intensity category. Categorical, total activity and weighted total activity scores are calculated.
Short Symptom Inventory | 2 months
  It is a 53-item multidimensional symptom screening scale developed by Derogatis (1992). It consists of 9 subscales and 3 global indexes. These; It includes somatization, obsessive-compulsive symptom, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid thought, and psychoticism dimensions. The scoring of the items is in the liker type between 0 and 4. The total score range varies between "0-212". It is evaluated that the higher the score, the higher the frequency of mental symptoms. Subscale scores are obtained by dividing the sum of the scores given to the items forming each subscale by the number of items.

SECONDARY OUTCOMES:
World Health Organization Quality of Life Scale Short Form (WHOQOL-BREF) | 2 months
  The scale evaluates physical, mental, social and environmental well-being and consists of 26 questions. Field scores range from 4 to 20, and the higher the score, the higher the quality of life.
Fatigue Severity Scale | 2 months
  The Scale is shown as the best example among one-dimensional scales. Each item of the scale, which consists of 9 items that patients can apply to themselves, is scored between 1-7 and the total score is calculated by taking the average of 9 items. The cut-off value for pathological fatigue was determined as 4 and above. The lower total scores mean less fatigue.
Pittsburgh Sleep Quality Index | 2 months
  The scale is a 19-item self-report scale that evaluates sleep quality and disturbance in the past month. It consists of 24 questions, 19 questions self-report questions, 5 questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use, and Daytime Dysfunction. Each component is evaluated over 0-3 points. The total score of the 7 components gives the scale total score. The total score ranges from 0 to 21. A total score greater than 5 indicates "poor sleep quality".

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat Yaprak Cetin, Asst Prof, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University Clinical Research Ethics Commitee, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No